CLINICAL TRIAL: NCT03254186
Title: Safety and Efficacy of Propranolol in the Treatment of Tardive Dyskinesia
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: No participants
Sponsor: Emory University (Other)
Collaborators: Atlanta Clinical and Translational Science Institute (Other)
Responsible Party: Principal Investigator, Jaime Hatcher-Martin, Asstant Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00096912
Record Dates: First submitted 2017-08-16; First posted 2017-08-18 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Tardive Dyskinesia
Keywords: Propranolol; Safety; Efficacy; Tardive Dyskinesia treatment
MeSH Terms: conditions — Tardive Dyskinesia | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propranolol Hydrochloride (Experimental): Two week up-titration to reach a total dose of 20mg per oral four times per day over the first two weeks then will remain on a stable dose for six weeks. The patients will be treated for eight weeks, complete a one week washout and then crossed over to another arm for eight weeks.
  Interventions: Drug: Propranolol Hydrochloride
- Placebo Oral Tablet (Placebo Comparator): Identical placebo. The patients will be treated for eight weeks, complete a one week washout and then crossed over to another arm for eight weeks.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Propranolol Hydrochloride — Propranolol is started 10 mg tablet twice per day per oral, two week up-titration to reach a total dose of 20mg per oral four times per day over the first two weeks, then will remain on a stable dose for six weeks.
  Other Names: Inderal
  Arms: Propranolol Hydrochloride
Drug: Placebo Oral Tablet — Identical placebo is started one tablet twice per day per oral, increase over the first two weeks to reach one tablet four times per day, then will remain on this dose for six weeks.
  Other Names: Placebo
  Arms: Placebo Oral Tablet

SUMMARY:
Tardive dyskinesia (TD) is a disabling, embarrassing and often irreversible iatrogenic movement disorder that can occur in anyone exposed to drugs that block dopamine receptors, including first and second generation antipsychotics and antiemetic agents. There is no way to prevent TD except preventing exposure to the inciting agents and there are no approved symptomatic therapies. Propranolol is an FDA-approved β-blocker with limited data supporting its use as a treatment for TD.

The goal of this study is to determine the efficacy of propranolol in the treatment of TD in a double-blind, cross-over prospective manner. If propranolol is found to be an effective therapy, it will fulfill a great need in the treatment of TD with a medication that is known to be safe and inexpensive.

DETAILED DESCRIPTION:
Tardive dyskinesia (TD) is a disabling, embarrassing and often irreversible iatrogenic movement disorder that can occur in anyone exposed to drugs that block dopamine receptors, including first and second generation antipsychotics and antiemetic agents. There is no way to prevent TD except preventing exposure to the inciting agents and there are no approved symptomatic therapies. Propranolol is an FDA-approved β-blocker with limited data supporting its use as a treatment for TD.

The goal of this study is to determine the efficacy of propranolol in the treatment of TD in a double-blind, cross-over prospective manner. Patients with a diagnosis of TD will be randomized to propranolol or identical placebo. The patients will be treated for eight weeks, complete a one week washout and then crossed over for another eight weeks. Hence, the subjects will be their own controls. Participation in this pilot trial will provide placebo controlled blinded data that will assist in planning a larger phase II trial. If propranolol is found to be an effective therapy, it will fulfill a great need in the treatment of TD with a medication that is known to be safe and inexpensive.

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 years
* diagnosis of classical TD by a movement disorder expert for at least 6 months with a baseline score of at least 2 on two of the seven items on the AIMS severity scale
* stable on medication (either on or off dopamine blocking agents) for at least six months.

Exclusion Criteria:

* breastfeeding
* pregnant
* unstable psychiatric disease
* history of asthma or COPD
* baseline heart rate less than 60
* history of orthostatic hypertension or its presence at screening
* history of congestive heart failure or unstable angina pectoris
* resting SBP <100 and DBP < 60
* AV-block II or III without pacemaker
* history of diabetes mellitus
* previous adverse effects from use of beta-blockers
* current use of a β-blocker and the other following drugs: quinidine, amiodarone, propafenone, digoxin, verapamil, diltiazem, clonidine, and warfarin
* tremor, dystonia, akathisia or other non-tardive movement disorder
* any medical illness that precludes treatment with propranolol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Change in the Abnormal Involuntary Movement Scale (AIMS) score. | Visit 1, 3 4, 6, 7 (up to 18 weeks)
  AIMS is a rating scale that scores each individual involuntary movement type at different body locations on a five-point anchored scale. For this study, items 1-7 represent the severity portion (rated 0-4) of the scale and will be used as the primary end point. This measure will be completed at the time of the visit by the enrolling physician. In addition, a standardized video documenting the motor portion of the AIMS will be completed at baseline and eight weeks for both segments of the study. These will be placed in a randomized order and scored using the AIMS severity scale by two blinded raters using consensus measures. A comparison of the change in score from placebo to active by the blinded video raters will be the primary outcome measure.

SECONDARY OUTCOMES:
Change in the Clinical Global Impression of Severity (CGI-S) score. | Visit 1, 3 4, 6 (up to 18 weeks)
  The CGI provides an overall clinician-determined summary measure that takes into account all available information, including a knowledge of the patient's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the patient's ability to function.
  The CGI-Severity (CGI-S) asks the clinician one question: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" which is rated on the following seven-point scale: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients.
  This rating is based upon observed and reported symptoms, behavior, and function in the past seven days. As symptoms and behavior can fluctuate over a week; the score should reflect the average severity level across the seven days.
Change in the Clinical Global Impression -Improvement (CGI-I) score. | Visit 3 and 6 (up to 18 weeks)
  The CGI-Improvement (CGI-I) is similarly simple in its format. Each time the patient is seen after medication has been initiated, the clinician compares the patient's overall clinical condition to the one week period just prior to the initiation of medication use (the so-called baseline visit). The CGI-I score obtained at the baseline (initiation) visit serves as a basis for making this assessment. Only the following one query is rated on a seven-point scale: "Compared to the patient's condition at admission to the project [prior to medication initiation], this patient's condition is: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment."

OTHER OUTCOMES:
Change in the Short Form-36 question health survey (SF-36v2) score. | Visit 1, 3 4, 6 (up to 18 weeks)
  The Short Form-36 question health survey (SF-36v2) measures a subject's functional health and well-being from their own point of view. SF-36v2 is comprised of 36 questions spanning eight health domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. The eight scaled scores are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. The health domain scales contribute to the scoring of two summary measures: physical health and mental health.
Change in the Craniocervical Dystonia Questionnaire (CDQ-24) score. | Visit 1, 3 4, 6 (up to 18 weeks)
  A modified version of the CDQ-24, a questionnaire to evaluate the quality of life in patients with face/neck movement disorders such as cervical dystonia and blepharospasm. The 24 questions of the CDQ-24 are divided in five areas:stigma (6), emotional wellbeing (5), pain (3), activities of daily living (6) and family/social life (4). Each question has five possible answers, in which 0 (zero) is the best and 4 is the worst. The total score of the CDQ-24 ranges from 0 (best Quality of Life) to 100 (worst Quality of Life).

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Hatcher-Martin, MD, PhD, Principal Investigator — Emory University

IPD SHARING:
Plan to Share IPD: Undecided